CLINICAL TRIAL: NCT04440592
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate Efficacy, Safety, and Tolerability of MT-7117 in Subjects With Diffuse Cutaneous Systemic Sclerosis
Brief Title: Study to Evaluate Efficacy, Safety, and Tolerability of MT-7117 in Subjects With Diffuse Cutaneous Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-7117-G02
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MT-7117 (Experimental): Oral tablet of MT-7117 once a day.
  Interventions: Drug: MT-7117
- Placebo (Placebo Comparator): Oral tablet of placebo once a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-7117 — MT-7117
  Other Names: Dersimelagon
  Arms: MT-7117
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of MT-7117 treatment in subjects with diffuse cutaneous systemic sclerosis (dcSSc) using the American College of Rheumatology Composite Response Index in Diffuse Systemic Sclerosis (ACR CRISS) at Week 52

ELIGIBILITY:
Additional screening criteria check may apply for qualification.

Inclusion Criteria:

* Subjects who meet all the following criteria will be considered eligible to participate in the study:

  1. Must provide signed and dated informed consent form (ICF) to participate in the study. Subjects must be able to (in the judgment of the Investigator) understand the nature of the study and all risks involved with participation in the study. Subjects must be willing to cooperate and comply with all protocol restrictions and procedures including study visits.
  2. Male or female age ≥ 18 years at screening with documented diagnosis of systemic sclerosis (SSc), as defined using the 2013 ACR/European League Against Rheumatism (EULAR) criteria.
  3. Has diffuse cutaneous form of SSc according to Leroy and Medsger's criteria.
  4. Disease duration ≤ 5 years from the first non-Raynaud's phenomenon manifestation.
  5. Has an mRSS of 15 to 45 units at screening and have clinical skin involvement proximal and distal to the elbows, knees, or both or any truncal involvement, with or without face involvement.
  6. If disease duration is > 24 months defined as time from the first non Raynaud phenomenon manifestation, subject must fulfill at least 1 of the criteria listed below that are indicatives of active disease at screening:

     1. A documentation of new skin involvement that occurred within the past 9 months, or
     2. Increase in mRSS ≥ 3 units within the past 9 months, or
     3. Presence of TFRs or,
     4. C- reactive protein (CRP) ≥ 6 mg/L, or
     5. Erythrocyte sedimentation rate ≥ 28 mm/hr, or
     6. Platelet count ≥ 330 x 10^9/L (330,000/microliter).

     NOTE: Investigator should exclude all other acute intercurrent illness if subjects fulfilling laboratory criteria (d, e, f) only.
  7. Willing to follow restrictions regarding concomitant medications that are described.
  8. Female subjects who are non-lactating and have a negative urine pregnancy test at baseline visit prior to receiving the first dose of study drug.
  9. Female subjects of childbearing potential and male subjects with partner of child-bearing potential currently using/willing to use 2 effective methods of contraception including barrier method as described.

Exclusion Criteria:

- Subjects will be excluded from the study if any of the following criteria apply:

1. Has a history or presence of rheumatic autoimmune diseases other than dcSSc unless the dominant features of the disease are dcSSc, as determined by the Investigator.
2. Has a pulmonary disease with FVC ≤ 50% of predicted at time of screening.
3. Has a diagnosis of clinically significant resting pulmonary hypertension (if exceeding estimated right ventricular systolic pressure of > 40 mmHg estimated by transthoracic echocardiography [unless the right heart catheterization is normal within the last 6 months] or mean pulmonary artery pressure > 30 mmHg as measured by right heart catheterization) and requires treatment with more than one oral medication.
4. Has a cardiac abnormality such as left ventricular failure with ejection fraction < 45%, significant arrhythmia, congestive heart failure (New York Heart Association Class II-IV), unstable angina, uncontrolled hypertension, or symptomatic pericardial effusion at screening.
5. Has a history of myocardial infarction in the last 26 weeks prior to screening.
6. Has a history of renal crisis within the past 52 weeks prior to screening.
7. Has a documented history of chronic kidney disease (stage 4-5, an estimated glomerular filtration rate [eGFR] < 30 mL/min at screening).
8. Presence or history of hepatobiliary disease at screening, determined as clinically significant by the Investigator after the discussion with the Sponsor Medical Monitor.
9. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) ≥ 2.0 × upper limit of normal (ULN), or total bilirubin > 1.5 × ULN at screening.
10. Has a history or presence of clinically significant disease not related to SSc [neurologic, renal, endocrinal, gastrointestinal cardiovascular, hepatic, dermatologic, hematological, musculoskeletal, genitourinary, thromboembolic, advanced arteriosclerosis, hyperthyroidism, moderate to severe hypertension, immunologic disease, pulmonary (e.g., uncontrolled asthma, emphysema, chronic obstructive pulmonary disease) or any other disorder] as determined by the Investigator at screening. Conditions deemed not-clinically significant according to the Investigator's discretion are acceptable.
11. Has a history or presence of psychiatric disease judged to be clinically significant by the Investigator and which may interfere with the study evaluation and/or safety of the subject.
12. Has any clinically significant disease or laboratory abnormality judged to be clinically significant by the Investigator and which may interfere with the study evaluation and/or safety of the subject at screening. Laboratory abnormalities include but not limited to any of the followings: Hemoglobin < 9 g/dL; WBC < 3,000/mm3 (< 3 x 10^9/L); platelets < 100,000/mm3 (<100 x 10^9/L).
13. Has a history of positive hepatitis B surface antigen, hepatitis C antibody, except for documented cure for the hepatitis B virus (HBV), defined as sustained, undetectable HBsAg and HBV DNA in serum and adequately treated hepatitis C virus (HCV) with documentation of sustained virologic response defined as undetectable HCV RNA at least 12 weeks after the end of treatment.
14. Has a history of positive human immunodeficiency virus (HIV)
15. Has a history of melanoma, familial melanoma (defined as having 2 or more first-degree relatives, such as parent, sibling, and/or child), or presence of melanoma and/or lesions suspicious for melanoma at screening.
16. Has a presence of squamous cell carcinoma, basal cell carcinoma, or other malignant skin lesions. Any suspicious lesions or nevi (Melanocytic Lesions) will be evaluated. If the suspicious lesion or nevi (Melanocytic Lesions) cannot be resolved through biopsy or excision, the subject will be excluded from the study.
17. Has history of any other malignancy(ies) in the last 5 years with the exception of cervical carcinoma in situ.
18. Has a history or planning to receive cell-depleting therapy or bone marrow transplantation during study treatment period.
19. Has a history of ultraviolet (UV) phototherapy within 6 weeks prior to screening or planning to receive UV phototherapy during study treatment period.
20. Treatment of SSc disease with

    1. Cyclophosphamide, rituximab, or cyclosporine received within 26 weeks prior to screening.
    2. Small molecules such as JAK inhibitors (e.g., tofacitinib) received within 12 weeks prior to screening.
    3. Pirfenidone received within 12 weeks prior to screening.
    4. Infliximab, certolizumab, golimumab, adalimumab, abatacept, tocilizumab within 10 weeks prior to screening.
    5. Etanercept within 4 weeks prior to screening.
    6. Oral, intravenous, or intramuscular corticosteroids (prednisone > 10 mg/day or equivalent) received within 30 days prior to screening
    7. Nintedanib within 12 weeks prior to screening.
    8. More than 1 of the immunosuppressant therapy listed below as concomitant therapy with study drug, has changed one of the medication below within 12 weeks prior to screening, or not on a stable dose of the same medication for at least 12 weeks prior to screening.

       * i. Mycophenolate (up to 3 g/day), or
       * ii. Mycophenolic acid (up to 2.14 g/day), or
       * iii. Methotrexate (up to 25 mg/Week), or
       * iv. Leflunomide (up to 20 mg/day), or
       * v. Azathioprine (up to 3 mg/kg/day).
21. Treatment with afamelanotide or other MC1R agonist within 12 weeks before screening (Visit 1).
22. Treatment with any drugs or supplements which, in the opinion of the Investigator, may interfere with the objectives of the study or safety of the subject.
23. Has previously exposed to MT 7117 (this does not include placebo treated subjects).
24. Has previously treated with any investigational agent within 12 weeks prior to screening OR 5 half-lives of the investigational product (whichever is longer).
25. Female subjects who are pregnant, lactating, or intending to become pregnant during the study.
26. Has a positive autoantibody status of anti-centromere antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (34):
- United States (11):
  - Arizona Arthritis, Glendale, Arizona
  - Pacific Arthritis Care Center, Los Angeles, California
  - The Board of Trustees of the Leland Stanford Junior University, Redwood City, California
  - Yale School of Medicine - The Anlyan Center (TAC) for Medical Research & Education, New Haven, Connecticut
  - GNP Research, Hollywood, Florida
  - Millennium Research, Ormond Beach, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Shelby Research, LLC, Memphis, Tennessee
  - The University of Texas Medical School at Houston, Houston, Texas
- Belgium (3):
  - UZ Leuven, Leuven, Vlaam Gewest
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Universitaire (CHU) de Liege - Domaine Universitaire du Sart Tilman, Liège
- Mount Sinai Hospital, The Rebecca Macdonald Centre For Arthritis And Autoimmune Disease, Toronto, Ontario, Canada
- Germany (3):
  - University Hospital Of Tuebingen, Tübingen, Baden-Wuettemberg
  - CIRI, Centrum fur innovative Diagnostik und Therapie Rheumatologie und Immunologie (GmbH) Am Klinikum der Johann Wolfgang Goethe-Universitat, Frankfurt am Main, Hesse
  - Internistisches Zentrum des Universitaetsklinikums Erlangen, Erlangen
- Italy (2):
  - University of Ferrara Azienda Ospedaliero-Universitaria Sant' Anna, Cona, Ferrera
  - Universita degli Studi di Milano - Azienda Ospedaliera Istituto Ortopedico Gaetano Pini, Milan, Lombardy
- Poland (7):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Centrum Kliniczno-Badawcze J.Brzezicki, B.Gornikiewicz-Brzezicka Lekarze Spolka partnerska, Elblag
  - Malopolskie Centrum Kliniczne, Krakow
  - Centrum Medyczne Plejady, Krakow
  - Medyczne Centrum Hetmanska, Poznan
  - Medycyna Kliniczna, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
- Spain (5):
  - Institut d'Investigacio i Innovacio Parc Tauli, Hospital Universitari Parc Taulí, Sabadell, Barcelona
  - Hospital Del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
- United Kingdom (2):
  - Western General Hospital, Edinburgh
  - The Royal Free Hospital - Royal Free London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ogasawara A, Ide R, Inoue S, Tsuda M, Teng R. Assessment of Potential Drug-Drug Interactions for Novel Oral Melanocortin-1 Receptor Agonist Dersimelagon. Pharmacol Res Perspect. 2025 Feb;13(1):e70069. doi: 10.1002/prp2.70069. PMID 39887900

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MT-7117 | Placebo
Started | 38 | 38
Completed | 28 | 36
Not Completed | 10 | 2
Not completed — Adverse Event | 8 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other therapy needed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MT-7117 | Placebo | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (12.5) | 54.2 (12.4) | 51.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 56
  Male | 12 | 8 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Non-hispanic or Latino | 31 | 29 | 60
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: The ACR CRISS Composite Score (0-1) at Week 52
Description: The comparison between MT-7117 treatment group and placebo group will be performed. The ACR CRISS exponential algorithm determines the predicted probability of improvement from baseline, incorporating change in mRSS, FVC % predicted, physician and patient global assessments, and HAQ-DI. The outcome is a continuous variable between 0.0 and 1.0 (0 - 100%). A higher score indicates greater improvement.
Time Frame: Week 52
Population: Reason of discrepancy between Number analyzed" and "Overall Number of Participants Analyzed: The analysis was performed only in patients who have data at week 52.
Measure: Median (Full Range); unit: scores on ascale
Arm/Group | MT-7117 | Placebo
Number analyzed (Participants) | 25 | 33
scores on ascale | 0.8537 [0.000 to 1.000] | 0.8502 [0.000 to 1.000]

2. Secondary Outcome: Change in Health Assessment Questionnaire Disability Index (HAQ-DI) From Baseline up to Week 52
Description: To evaluate the efficacy of MT 7117 treatment for up to 52 weeks using the Health Assessment Questionnaire Disability Index (HAQ DI). The Health Assessment Questionnaire Disability Index (HAQ-DI) is a self-administered instrument consists of 20 questions referring to eight component sets consisting of dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Each item is scored on a 4-point scale from 0 to 3: 0 = Without any difficulty; 1 = With some difficulty; 2 = With much difficulty; 3 = Unable to do. Overall score was computed as the sum of component set scores and divided by the number of component sets answered. This outcome measure represents the change in mean score from baseline. A negative change from baseline indicates improvement.
Time Frame: 52 weeks
Population: The analysis was performed only in patients who have data at each week.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MT-7117 | Placebo
Number analyzed (Participants) | 33 | 38
score on a scale
  Change from baseline (BL) at Week 16 | -0.1439 (0.3803) | -0.0395 (0.3900)
  Change from BL at Week 26: number analyzed (Participants) | 31 | 38
  Change from BL at Week 26 | -0.0847 (0.3360) | -0.0691 (0.4481)
  Change from BL at Week 39: number analyzed (Participants) | 31 | 37
  Change from BL at Week 39 | -0.0927 (0.3178) | -0.0439 (0.5147)
  Change from BL at Week 52: number analyzed (Participants) | 27 | 36
  Change from BL at Week 52 | -0.1111 (0.4265) | -0.0208 (0.5102)

3. Secondary Outcome: Change in Percent Predicted Forced Vital Capacity (%pFVC) From Baseline up to Week 52
Description: To evaluate the efficacy of MT-7117 treatment for up to 52 weeks on pulmonary function as measured by percent predicted forced vital capacity (%pFVC)
Time Frame: 52 weeks
Population: Reason of discrepancy between Number analyzed" of each row and "Overall Number of Participants Analyzed": The analysis was performed only in patients who have data at each week.
Measure: Mean (Standard Deviation); unit: %pFVC
Arm/Group | MT-7117 | Placebo
Number analyzed (Participants) | 30 | 35
%pFVC
  Change from BL at Week 16 | 0.754 (4.938) | -1.058 (5.749)
  Change from BL at Week 26: number analyzed (Participants) | 28 | 35
  Change from BL at Week 26 | 0.904 (5.669) | -0.691 (5.847)
  Change from BL at Week 39: number analyzed (Participants) | 30 | 34
  Change from BL at Week 39 | -1.201 (6.293) | -1.457 (5.600)
  Change from BL at Week 52: number analyzed (Participants) | 26 | 33
  Change from BL at Week 52 | 0.048 (6.917) | -2.906 (5.101)

4. Secondary Outcome: Change in Patient Global Assessment From Baseline up to Week 52
Description: To evaluate the efficacy of MT-7117 treatment for up to 52 weeks using the Patient Global Assessment
Time Frame: 52 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MT-7117 | Placebo
Number analyzed (Participants) | 34 | 38
score on a scale
  Change from BL at Week 16 | -0.8 (1.8) | -0.3 (1.9)
  Change from BL at Week 26: number analyzed (Participants) | 32 | 38
  Change from BL at Week 26 | 0.0 (2.5) | -0.4 (2.6)
  Change from BL at Week 39: number analyzed (Participants) | 32 | 37
  Change from BL at Week 39 | -0.7 (2.2) | -0.5 (2.3)
  Change from BL at Week 52: number analyzed (Participants) | 28 | 36
  Change from BL at Week 52 | -0.5 (2.3) | -0.3 (2.5)

5. Secondary Outcome: Change in Physician Global Assessment From Baseline up to Week 52
Description: To evaluate the efficacy of MT-7117 treatment for up to 52 weeks using the Physician Global Assessment. The Physician Global Assessment is used to assess the physician's rating of overall health of the subject. Physicians rate the perceived health of the subject on an 11-point scale from 0 (excellent) to 10 (extremely poor).
Time Frame: 52 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MT-7117 | Placebo
Number analyzed (Participants) | 34 | 38
score on a scale
  Change from BL at Week 16 | -1.6 (1.9) | -1.7 (1.8)
  Change from BL at Week 26: number analyzed (Participants) | 32 | 38
  Change from BL at Week 26 | -1.6 (2.1) | -1.7 (2.1)
  Change from BL at Week 39: number analyzed (Participants) | 32 | 37
  Change from BL at Week 39 | -2.1 (2.5) | -2.2 (2.3)
  Change from BL at Week 52: number analyzed (Participants) | 28 | 36
  Change from BL at Week 52 | -2.0 (2.9) | -1.7 (2.2)

6. Secondary Outcome: Change in Modified Rodnan Skin Score (mRSS) From Baseline From Baseline up to Week 52
Description: To evaluate the efficacy of MT-7117 treatment for up to 52 weeks using the modified Rodnan Skin Score (mRSS). mRSS evaluates a subject's skin thickness which will be assessed by palpation and rated using an mRSS that ranges from 0 (normal) to 3 (severe skin thickening) across 17 different body sites. The total score is the sum of the individual skin scores from all of these sites and ranges from 0 to 51 units.
Time Frame: 52 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MT-7117 | Placebo
Number analyzed (Participants) | 34 | 38
score on a scale
  Change from BL at Week 16 | -3.2 (4.7) | -3.6 (3.9)
  Change from BL at Week 26: number analyzed (Participants) | 32 | 37
  Change from BL at Week 26 | -4.9 (5.5) | -5.3 (6.9)
  Change from BL at Week 39: number analyzed (Participants) | 32 | 36
  Change from BL at Week 39 | -6.4 (7.0) | -6.2 (7.5)
  Change from BL at Week 52: number analyzed (Participants) | 28 | 36
  Change from BL at Week 52 | -6.6 (8.2) | -6.5 (7.9)

7. Secondary Outcome: ACR CRISS Score up to Week 39
Description: To evaluate the efficacy of MT 7117 treatment for up to 39 weeks using the ACR CRISS Score. The ACR CRISS exponential algorithm determines the predicted probability of improvement from baseline, incorporating change in mRSS, FVC % predicted, physician and patient global assessments, and HAQ-DI. The outcome is a continuous variable between 0.0 and 1.0 (0 - 100%). A higher score indicates greater improvement.
Time Frame: 39 weeks
Population: as for outcome 3
Measure: Median (Full Range); unit: scores on ascale
Arm/Group | MT-7117 | Placebo
Number analyzed (Participants) | 29 | 35
scores on ascale
  Week 16 | 0.0349 [0.000 to 1.000] | 0.1236 [0.000 to 1.000]
  Week 26: number analyzed (Participants) | 28 | 34
  Week 26 | 0.2626 [0.000 to 1.000] | 0.6232 [0.000 to 1.000]
  Week 39: number analyzed (Participants) | 29 | 33
  Week 39 | 0.3890 [0.000 to 1.000] | 0.5289 [0.000 to 1.000]

8. Secondary Outcome: ACR CRISS Score Responder (CRISS>=0.6) From Baseline up to Week 52
Description: To evaluate the efficacy of MT-7117 treatment for up to 52 weeks using CRISS Score. Subjects with CRISS score is >=0.60 are considered improved, while subjects with CRISS score < 0.60 are considered not improved.
Time Frame: 52 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | MT-7117 | Placebo
Number analyzed (Participants) | 29 | 35
Participants
  Week 16 | 10 | 8
  Week 26: number analyzed (Participants) | 28 | 34
  Week 26 | 10 | 18
  Week 39: number analyzed (Participants) | 29 | 33
  Week 39 | 11 | 15
  Week 52: number analyzed (Participants) | 25 | 33
  Week 52 | 14 | 18

ADVERSE EVENTS:
Time Frame: 60 weeks
Arm/Group | MT-7117 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 4/38 | 2/38
Other Adverse Events (participants affected / at risk) | 35/38 | 28/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-7117 (N=38) | Placebo (N=38)
Pneumonia (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MT-7117 (N=38) | Placebo (N=38)
Cataract (Eye disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 10 | 5
Dysphagia (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 7 | 2
Vomiting (Gastrointestinal disorders) | 6 | 2
Fatigue (General disorders) | 4 | 3
Bronchitis (Infections and infestations) | 2 | 1
COVID-19 (Infections and infestations) | 4 | 5
Gastroenteritis (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 2
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 2
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Headache (Nervous system disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Nail pigmentation (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 8 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 16 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Solar lentigo (Skin and subcutaneous tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT04440592/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT04440592/SAP_001.pdf